CLINICAL TRIAL: NCT03466879
Title: A User Study of SYNUS Pain Relief Made by Tivic Health Systems
Status: Completed | Type: Observational
Sponsor: Tivic Health Systems (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: CP00001
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Sinus; Inflammation
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Active device users: Users will use an active SYNUS Pain Relief device
  Interventions: Device: SYNUS Pain Relief device
- Sham device users: Users will use a sham SYNUS Pain Relief device that is not providing treatment

INTERVENTIONS:
Device: SYNUS Pain Relief device — SYNUS Pain Relief is a handheld micro-current TENS device used for the temporary relief of sinus pain.
  Groups: Active device users

SUMMARY:
Demonstrate the ability of subjects suffering from sinus pain to self-treat with the SYNUS Pain Relief device and to obtain pain relief compared to a sham/placebo device.

DETAILED DESCRIPTION:
A prospective study of at least 58 recruited subjects suffering from sinus pain. At least 30 of the subjects will be randomly selected to use the SYNUS Pain Relief device, a device that uses micro-currents to stimulate major nerve fibers passing from the sinus passages through various foramina to the facial skin. Subjects will read manufacturer's provided Instructions-For-Use (IFU's) and without help from staff will proceed to self-perform the treatment. The other subjects will follow the same procedure but use a sham/placebo device with no stimulating current. Subjects will be blinded as to the device they use. Prior to and 10 minutes following the stimulation, subjects will score their pain level on a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age and older
* Present with symptoms of sinus pain and pressure
* Have an initial sinus pain score of 4 or more on the visual analogue scale
* Be able to read and understand English
* Agree to participate in the study
* Be able and willing to provide Informed Consent

Exclusion Criteria:

* Do not meet Inclusion Criteria
* Have currently a dental infection
* Have currently abnormal cranial nerve or other neurological findings or symptoms that would require prompt medical attention
* Be currently pregnant
* Have implanted electrostimulation devices including a pacemaker, a DBS or a cochlear implant

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At least 58 subjects suffering from sinus pain
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 10 minutes
  Average decrease in pain score of the SYNUS device is greater than the average decrease is pain score for the sham/placebo device.

CONTACTS AND LOCATIONS:
Overall Officials: Jayakar Nayak, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No